CLINICAL TRIAL: NCT02507739
Title: Evaluation of the Impact of an Outpatient Obstetric Epidurals During Labor
Acronym: PERIAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-097
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Obstetric Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- possibility to walk during labor (Other): possibility to walk during labor
  Interventions: Other: possibility to walk during labor
- no possibility to walk during labor (Other): no possibility to walk during labor
  Interventions: Other: no possibility to walk during labor

INTERVENTIONS:
Other: no possibility to walk during labor
  Arms: no possibility to walk during labor
Other: possibility to walk during labor
  Arms: possibility to walk during labor

SUMMARY:
Mobilization, ambulation, during obstetrical work attitudes are naturally adopted by women since ancient times in many countries. The advent of the epidural in the 60s revolutionized the management of pain during childbirth. The consideration of such advance is to keep the laboring parturients lying down. Indeed at this time the use of high doses of local anesthetics charge of an engine block against formally allocate all up.

In a matchless analgesic efficacy during childbirth, epidurals also offers the possibility of a secure obstetrical gesture because without general anesthesia, inhalation great purveyor in these women with full stomach. These advantages explain the considerable growth in the number of epidurals performed in obstetric work in France over the last thirty years. However, this analgesia technique will soon be implicated in the alterations of obstetric mechanics, its effects depend primarily on the nature and concentration of the products used.

Evolution is then marked by a considerable reduction of concentrations of local anesthetics used with the addition of opioids, allowing to achieve an isolated analgesia without impairing motor skills, it involves the lower limbs or muscles pelvis, allowing the woman to mobilize.

Ambulatory epidural and made its appearance in the early 90. Responding to women in labor demand wishing to receive effective labor analgesia without being confined to bed, she then puts to the test the dogmas and practices on how to provide analgesia that is both effective and safe. It is now well codified and used daily in some maternity hospitals.

The mobilization of women during labor is a subject that motivates obstetric teams Caen University Hospital for many years. Motherhood has thus given the means for monitoring and ambulatory epidural analgesia protocol suitable for this technique.

The introduction of this daily care protocol opens new possibilities of care delivery hoped more physiological and less iatrogenic.

A critical evaluation of the changes possibly recorded on obstetric mechanics inherent question, motivating, for which the answers are now few and discordant in the literature.

The investigators therefore propose a randomized study evaluating single-center relative to obstetrical work typically occurring in a bed, the mobilizations of repercussions out of bed, in terms of obstetrical mechanics and comfort of the parturient.

Those will be objectified by a significant change in the working hours. This study included 560 patients is scheduled to last 2 years. Positive effects could also have repercussions in terms of public health and even of health economics.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman Over 18 years, beneficiary of social security / CMU
* pregnant woman Receiving the newsletter and do not express opposition.
* pregnant woman of More than 35 weeks of amenorhea, admitted to the start of work or for inducing labor
* Fetus in cephalic presentation
* pregnant woman Under ANALGESIA EPIDURAL (0.0625% levobupivacaine protocol CHU Caen)

Exclusion Criteria:

* refusal by the patient
* multiple pregnancy
* see, polyhydramnios
* unbalanced gestational hypertension, pre-eclampsia
* prematurity <35 SA
* retard Intra uterine growth
* fetal Malformations
* need Internal tocometry, but especially a recording FHR intrauterine route (electrode scalp)
* RCF insufficient (<80%)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
labor time | baseline